CLINICAL TRIAL: NCT05978986
Title: Efficiency of Determining the Clinical Class of Chronic Venous Disorders by Artificial Intelligence (IVENUS App)
Brief Title: Efficiency of Determining the Clinical Class of Chronic Venous Disorders by Artificial Intelligence
Acronym: IVENUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinic of Phlebology and Laser Surgery, Chelyabinsk, Russia (Other)
Responsible Party: Principal Investigator, Denis Borsuk, Director, Clinic of Phlebology and Laser Surgery, Chelyabinsk, Russia
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: 17122021
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Varicose Veins of Lower Limb; Telangiectasia
MeSH Terms: conditions — Telangiectasis

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Determining of the clinical class of chronic venous disorders by artificial intelligence — The doctor takes pictures of the lower extremities and uploads them to the IVENUS application, which automatically determines the clinical class according to CEAP. Further, the doctor independently determines the clinical class according to CEAP and enters the data into the register.

SUMMARY:
Purpose: To evaluate the sensitivity and specificity of the method for determining the clinical class of chronic venous diseases using the Ivenus application (within C0-C2 according to CEAP).

Materials and methods: Patients who applied to several phlebology clinics for an initial consultation are consistently included in a multicenter prospective study. At the appointment, a doctor with at least 5 years of experience takes photographs of the lower extremities and uploads them to the IVENUS application, which automatically determines the clinical class according to CEAP, without showing the results to the surgeon (blinding). Further, the doctor independently determines the clinical class according to CEAP and enters the data into the register.

The object of the study is a photograph of a certain area of the lower limb.

ELIGIBILITY:
Inclusion Criteria:

* C0-C2 CEAP clinical class;
* Signed consent to take part in investigation.

Exclusion Criteria:

* C3-C6 CEAP clinical class;
* Skin diseases of the lower extremities;
* Immobilization.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1530 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Determination of the sensitivity and specificity | 1 day
  Determination of the sensitivity and specificity of the method for determining the clinical class of chronic venous diseases according to the CEAP classification using the IVENUS application (within C0-C2 classes).

SECONDARY OUTCOMES:
Number of participants with complications | 1 day
  Any serious adverse event will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Denis Borsuk, Study Chair — VenoClinica, "Vasculab" ltd.
Locations (3):
- Russia (3):
  - Phlebolog ltd., Perm
  - Azbuka zdoroviya ltd., Yekaterinburg
  - Vasculab ltd., Yekaterinburg

IPD SHARING:
Plan to Share IPD: No